CLINICAL TRIAL: NCT06437457
Title: Comparison of CE-MRI and CEUS for Measuring Tumor Size of HCC
Brief Title: Comparison of Gd-EOB-DTPA-enhanced MRI and Contrast-enhanced Ultrasound for Measuring Tumor Size of Solitary Hepatocellular Carcinoma ≤ 5cm:A Retrospective Study
Status: Completed | Type: Observational
Sponsor: Anhui Medical University (Other)
Responsible Party: Principal Investigator, Kunyuan Jiang, Anhui Medical University, Anhui Medical University
Other Study IDs: 2023-RE-117
Record Dates: First submitted 2024-05-25; First posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: HCC - Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CEUS: The patients who underwent CEUS before liver resection
  Interventions: Radiation: ceus
- CE-MRI: The patients who underwent CE-MRI before liver resection
  Interventions: Radiation: ceus

INTERVENTIONS:
Radiation: ceus — MRI was performed by using a superconducting magnet scanner operated at 3.0 T (GE discovery MR750w, USA) and the CEUS examination (Mindray, China), ultrasound was performed first in B-mode to identify the suspicious lesions and then switched to contrast mode prior to the injection of the contrast medium.

SUMMARY:
Knowing the tumor size before operation is of great significance to the choice of treatment methods of surgeons and the prognosis of patients. In this study, two commonly used imaging methods( CE-MRI/CEUS) were selected to measure and compare the tumor size before operation, in order to determine which measurement method is more accurate.

DETAILED DESCRIPTION:
A total of 194 patients who met the inclusion criteria from January 2019 through May 2024 were included. Taken pathological results as the gold standard, Paired T-test and Bland-Altman analisis were conducted to assess the correlation and mean absolute error between the measured tumor sizes obtained from CE-MRI/CEUS and pathological results.

ELIGIBILITY:
Inclusion Criteria:

1. had no anti-HCC therapy before imaging examinations.
2. at least had one examination of Gd-EOB-DTPA-enhanced MRI and CEUS 2 weeks before surgery and confirmed as one single HCC.
3. If the patient had both imaging tests, the time interval between two examinations was less than 1 weeks.
4. both radiological and pathological results recorded the maximum tumor diameter.

Exclusion Criteria:

1. had anti-HCC therapy before imaging examinations.
2. had no examination of Gd-EOB-DTPA-enhanced MRI or CEUS 2 weeks before surgery .
3. had no radiological or pathological results recorded the maximum tumor diameter.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients who underwent liver resection from January 2019 to May 2024 were included.
Sampling Method: Non-Probability Sample
Enrollment: 194 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-20 (Actual)

PRIMARY OUTCOMES:
measuring HCC diameter | Jaunary 2019 - May 2024
  the performance of Gd-EOB-DTPA-enhanced MRI (CE-MRI) and Contrast-enhanced Ultrasound (CEUS) in measuring tumor size of solitary hepatocellular carcinoma (HCC) ≤5cm.

CONTACTS AND LOCATIONS:
Locations (1):
- Anhui Provincial Hospital, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: Undecided